CLINICAL TRIAL: NCT01847664
Title: A Randomised, Double-blind, Double-dummy, Multi-centre, Comparative Parallel-group Study to Evaluate the Efficacy of Oral Rifamycin SV-MMX® 400 mg b.i.d. vs. Rifamycin SV-MMX® 600 mg t.i.d. vs. Placebo in the Treatment of Acute Uncomplicated Diverticulitis
Brief Title: Rifamycin SV-MMX® 400 mg b.i.d. vs. Rifamycin SV-MMX® 600 mg t.i.d. vs. Placebo in Acute Uncomplicated Diverticulitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dr. Falk Pharma GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RIT-4/DIV
Record Dates: First submitted 2013-04-26; First posted 2013-05-07 (Estimated); Last update posted 2017-07-26 (Actual); Status verified 2017-07

CONDITIONS: Uncomplicated Diverticulitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Rifamycin SV-MMX® 400 mg b.i.d. (Experimental): Rifamycin SV-MMX® 800 mg
  Interventions: Drug: Rifamycin SV-MMX® 400 mg b.i.d.
- Rifamycin SV-MMX® 600 mg t.i.d. (Experimental): Rifamycin SV-MMX® 1800 mg
  Interventions: Drug: Rifamycin SV-MMX® 600 mg t.i.d.
- Rifamycin SV-MMX® Placebo (Placebo Comparator): Rifamycin SV-MMX® placebo
  Interventions: Drug: Rifamycin SV-MMX® Placebo

INTERVENTIONS:
Drug: Rifamycin SV-MMX® 400 mg b.i.d.
  Arms: Rifamycin SV-MMX® 400 mg b.i.d.
Drug: Rifamycin SV-MMX® 600 mg t.i.d.
  Arms: Rifamycin SV-MMX® 600 mg t.i.d.
Drug: Rifamycin SV-MMX® Placebo
  Arms: Rifamycin SV-MMX® Placebo

SUMMARY:
The purpose of the trial is to compare the efficacy of Rifamycin SV-MMX® 400 mg b.i.d. vs. Rifamycin SV-MMX® 600 mg t.i.d. vs. placebo in patients with acute uncomplicated diverticulitis.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent,
2. Patient is eligible for out-patient treatment,
3. Men or women between 18 and 80 years of age,
4. Diagnosis of left-sided uncomplicated diverticulitis confirmed by ultrasonography (US) and/or computed tomography (CT) according to modified Hinchey classification (stage 1a) or Hansen/Stock classification (stage I/IIa) or Ambrosetti classification (stage mild),
5. Presence of significant left lower quadrant pain during the last 24 hours before baseline,
6. CRP > ULN and/or leucocytosis (> ULN) at screening visit

Exclusion Criteria:

1. Existing complications of diverticulitis (diverticulitis with associated abscess, fistula, obstruction or perforation),
2. Right-sided diverticulitis,
3. Previous colonic surgery (except appendectomy, haemorrhoidectomy, and endoscopic removal of polyps),
4. Chronic inflammatory bowel disease (such as Crohn's disease, ulcerative colitis) or celiac disease,
5. Presence of symptomatic organic disease of the gastrointestinal tract (with the exception of non-bleeding hemorrhoids or hiatal hernia),
6. Hemorrhagic diathesis,
7. Active peptic ulcer disease,
8. Abnormal hepatic function or liver cirrhosis,
9. Abnormal renal function,
10. Colorectal cancer or a history of colorectal cancer,

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2013-08; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Rate of patients with treatment success at the day 10 visit | 10 days
  Treatment success includes e.g.:
  * absence of diverticulitis related symptoms
  * no complications of acute diverticulitis
  * no hospitalisation due to acute diverticulitis

SECONDARY OUTCOMES:
First visit with treatment success | 10 days
Rate of surgical intervention of acute diverticulitis | 10 days
Rate of hospitalisation due to acute diverticulitis | 10 days
Rate of occurrence of complicated diverticulitis | 10 days

CONTACTS AND LOCATIONS:
Locations (1):
- Evangelisches Krankenhaus Kalk, Cologne, North Rhine-Westphalia, Germany